CLINICAL TRIAL: NCT00099957
Title: A Clinical Study to Assess the Effect of Vildagliptin on Postprandial Lipid Parameters in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2217
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This study was not conducted in the United States. Many people with type 2 diabetes also have high cholesterol levels. The purpose of this study was to evaluate the effects of vildagliptin, an unapproved drug, on blood lipid measures such as triglycerides and cholesterol in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Genetic markers associated with increased risk of cardiovascular disease
* Not currently on drug therapy for type 2 diabetes
* Body mass index (BMI) in the range 25-40

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* High cholesterol as defined by the protocol
* Evidence of serious diabetic complications
* Other protocol-defined exclusion criteria may apply

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2003-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Postprandial serum total triglycerides at 4 weeks

SECONDARY OUTCOMES:
Postprandial total cholesterol at 4 weeks
Postprandial total apo B at 4 weeks
Postprandial triglycerides in the two lipoprotein fractions - chylomicrons and VLDL1+VLDL2+IDL (VLDL/IDL) at 4 weeks
Postprandial cholesterol in the two lipoprotein fractions - chylomicrons and VLDL1+VLDL2+IDL (VLDL/IDL) at 4 weeks
Postprandial apo B-48 and apo B-100 in the two lipoprotein fractions - chylomicrons and VLDL1+VLDL2+IDL (VLDL/IDL) at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland